CLINICAL TRIAL: NCT00253981
Title: Monochromatic Near-Infrared Light Energy (MIRE) in the Treatment of Tibial Stress Reaction
Brief Title: Light Therapy in the Treatment of Leg Pain
Acronym: MilCAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment not achieved succesfully
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WBAMC #05/13; CIRO #2005705 (Other: CIRO #2005705); NCT00253981 (Other Grant/Funding Number: NCT00253981)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Tibial Fractures; Leg Injuries
Keywords: Pain, Intractable; Infrared Rays; Leg
MeSH Terms: conditions — Tibial Fractures; Leg Injuries; Pain, Intractable

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infrared Light Therapy (Experimental): Intervention: The use of infrared light therapy for the treatment of tibial fracture. The treatment was assigned three times a week for four weeks.
  Interventions: Device: Monochromatic Near-Infrared Light Energy (MIRE)
- Standard of Care (Placebo Comparator): Standard of care was characterized by the use of standard medical treatment to include medication.
  Interventions: Device: Monochromatic Near-Infrared Light Energy (MIRE)

INTERVENTIONS:
Device: Monochromatic Near-Infrared Light Energy (MIRE) — Subjects randomized to the intervention group (Monochromatic Near-Infrared Light Energy), received treatment three times a week for a total of four weeks.

SUMMARY:
The purpose of this study is to apply Anodyne therapy to active duty soldiers, who have shin splints, to evaluate healing time and effectiveness.

DETAILED DESCRIPTION:
Tibial stress reactions and fractures are often difficult to treat, and therefore, many soldiers proceed to a medical disability/discharge. It is felt that with the use of the MIRE technology, active duty soldiers with tibial stress reactions and fractures will heal more quickly and completely. All soldiers will have a documented bone scintigraph as evidence for tibial stress reaction or fracture prior to enrollment. In addition, pain-pressure goniometric measures and time to complete the Balke protocol will also be used to assess healing with the MIRE technology.

Comparison: Soldiers with Active MIRE technology, compared to soldiers with Placebo MIRE technology.

ELIGIBILITY:
Inclusion Criteria:

* Active duty soldier
* Exertional leg pain of greater than 3 months duration
* Documented bone scintigraphic evidence for tibial stress reaction or fracture

Exclusion Criteria:

* Known leg Pathology other than stress reaction or fracture
* Service members known to be leaving area within next 6 months
* Pregnant females
* High risk cardiopulmonary patients
* Patients with assisted walking devices
* Patients with two or more cardiac risk factors

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LTC Richard P Petri, MD, Principal Investigator — Department of the Army
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment took place between 2006-2007 at a military treatment facility.
Pre-assignment Details: Some participants were excluded due to deployment, military training that required them to leave the post.
Period: Overall Study
Arm/Group | Infrared Light Therapy | Standard of Care
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: The experimental group received the monochromatic light infrared energy treatment (MIRE).
- Control: The control group followed the standard of care for the treatment of shin splints, usually physical therapy and medication.
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Numeric scale based on pain level (1-10). The higher the numeric value, the higher the pain level, as perceived by the participant.
Time Frame: 4 weeks
Arm/Group | Infrared Light Therapy | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Experimental: The experimental group received the monochromatic light infrared red energy treatment (MIRE).
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No